CLINICAL TRIAL: NCT05949359
Title: Effects of a Balance and Muscle Strengthening Exercise Program Using the Nintendo RingFit in Community-dwelling Older Adults With a History of Falls - a Feasibility Randomized Controlled Trial
Brief Title: The Feasibility of Nintendo RingFit to Improve Balance and Muscle Strength of Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URIS2021-111
Record Dates: First submitted 2023-07-09; First posted 2023-07-18 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Accidental Falls
Keywords: Falls; Exergaming; Feasibility studies; Aged

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nintendo RingFit exercise group (Experimental): Participants in the Nintendo RingFit exercise group received an 8-week, twice-weekly exercise program focusing on improving balance and lower limb muscle strength using Nintendo RingFit device.
  Interventions: Other: Nintendo RingFit-augmented exercise program
- Control group (No Intervention): Usual care was received by the control group participants.

INTERVENTIONS:
Other: Nintendo RingFit-augmented exercise program — Participants in the NRE group received an 8-week exercise training program using the Nintendo RingFit (60 minutes for each session, two sessions a week). In each session, the participants first performed 5 minutes of walk-up exercises (i.e., simple jogging), followed by 50 minutes of Nintendo RingFit exercises and 5 minutes of cool down exercises.
  The exercise intensity, in terms of repetitions, holding time of the exercise and advancement to difficult tasks, progressed gradually in 8 weeks.
  Arms: Nintendo RingFit exercise group

SUMMARY:
Background Existing findings have suggested that exergaming (i.e., exercise that requires people to move their body to play, providing an active gaming experience while serving as a form of physical activity), may have a potential to improve muscle strength and balance in older adults. However, no study has been conducted to investigate the effects of the Nintendo RingFit - an action role-playing game that aims to provide exercise training using a ring-shaped force sensor - in improving muscle strength and balance and possibly reducing falls in older adults living in the community.

Objective This study aims to investigate the feasibility of an exercise training program using Nintendo RingFit to improve balance and muscle strength among community-dwelling older adults.

Design A single-blind, randomized controlled feasibility trial.

Methods 30 participants will be recruited at local community-based elderly centers. Participants will be randomized to either the Nintendo RingFit-based exercise training group (NRE) or control group (CON) group with an allocation ratio of 1:1 by a researcher who will not participate in the recruitment and outcome evaluation. The NRE group will received an 8-week exercise training focusing on balance and lower limb muscle strength using the Nintendo RingFit. The CON group will receive a booklet and verbal instructions on the exercise for falls prevention, will be invited to join a leisure activity program (e.g., singing group) without any active exercise component for 8 weeks.

Outcomes The feasibility, acceptability and safety of the program will be examined at the end of the intervention. Postural balance, lower extremity strength, mobility, attention and executive function, fear of falling, and falls incidence of the participants will be assessed at 8 weeks.

Statistical analyses Descriptive statistics were presented for all variables. Chi-Square Test will be used to compare the difference in the proportion of fallers between the NRE and CON groups. Mann-Whitney U Test will be used to compare the functional outcomes between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* were 60 years old or above;
* had at least one fall in the past year;
* were able to walk independently without a walking aid for at least 10 meters;
* had no previous experience of using the Nintendo RingFit.

Exclusion Criteria:

* had a severe musculoskeletal, cardiopulmonary or neurological condition that limited their participation in the exercise program or assessment;
* had a significant visual or hearing impairment that limited their ability to follow exercise instructions;
* scored 18 or below in the Montreal Cognitive Assessment Hong Kong version (HK-MoCA) 4; or
* participated in any structured exercise program in the past 6 months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Adherence | Throughout the 8-week exercise program
  The attendance and retention of the participants in the trial
Adverse events | Throughout the 8-week exercise program
  The number of adverse events as a result of the exercise program
Acceptability | At 8-week post-intervention
  The acceptability of the participants toward the exercise program

SECONDARY OUTCOMES:
Mini-Balance Evaluation Systems Test | Week 0 (baseline) and week 8 (post-assessment)
  Balance, score range: 0 - 28, a higher score indicates better balance
Five-time-sit-to-stand test | Week 0 (baseline) and week 8 (post-assessment)
  Lower limb muscle strength, sec
Timed-Up and Go test - single and dual tasks | Week 0 (baseline) and week 8 (post-assessment)
  General mobility and dual task ability, sec
Iconographical Falls Efficacy Scale | Week 0 (baseline) and week 8 (post-assessment)
  Fear of falling, score range: 10 - 40, a higher score indicates greater fear of falling
Color Trails Test | Week 0 (baseline) and week 8 (post-assessment)
  Attention and executive function, sec

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No